CLINICAL TRIAL: NCT03267498
Title: Nivolumab in Combination With Chemoradiation for Patients With Stage II-IVB Nasopharyngeal Carcinoma, A Phase II Study With Correlative Biomarkers
Brief Title: Nivolumab + Chemoradiation in Stage II-IVB Nasopharyngeal Carcinoma (NPC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sue Yom (Other)
Collaborators: National University of Singapore (Other); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Sue Yom, Principal Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 162010; NCI-2017-02291 (Other: Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2017-08-23; First posted 2017-08-30 (Actual); Results first posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Nivolumab; Cisplatin; Radiotherapy

STUDY DESIGN:
Intervention Model Description: Single-arm, open label clinical trial of concurrent and adjuvant nivolumab, including a run-in phase to establish basic feasibility of the nivolumab schedule followed by expansion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nivolumab + chemoradiation (Experimental): Patients receive nivolumab IV over 60 minutes on day 1 of courses 1-5 and 7-12. Treatment repeats every 14 days for 11 courses in the absence of disease progression or unacceptable toxicity. Beginning at course 2, patients undergo radiation therapy QD 5 days per week and receive cisplatin IV over 30-60 minutes on day 1. Treatment repeats every 7 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Nivolumab; Drug: Cisplatin; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Nivolumab — Dosage 240mg of Nivolumab will be given intravenously over 60 minutes, every 14 days.
  Other Names: Opdivo
Drug: Cisplatin — Dosage 40 mg/m2 of cisplatin will be given intravenously over 30-60 minutes, every 7 days.
Radiation: Radiation Therapy — 2.12 Gy/fraction x 33 fractions of radiation therapy will be given, daily Monday - Friday

SUMMARY:
This phase II trial studies how well nivolumab and chemoradiotherapy works in treating patients with stage II-IVB nasopharyngeal cancer. Monoclonal antibodies, such as nivolumab, may block tumor growth in different ways by targeting certain cells. Chemoradiotherapy is the combination of chemotherapy and radiation therapy and may prevent the cancer from spreading when combined with nivolumab. Giving nivolumab and chemoradiotherapy may work better in treating patients with stage II-IVB nasopharyngeal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish the feasibility of treatment completion of a combined chemoradiation-nivolumab regimen followed by adjuvant nivolumab.

SECONDARY OBJECTIVES:

I. To determine the overall response rate at 1 year from end of treatment, as determined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria.

II. To determine the locoregional control rate at 1 year post-treatment.

III. To determine the distant metastasis rate at 1 year post-treatment.

IV. To determine the rate of Epstein-Barr virus (EBV) deoxyribonucleic acid (DNA) clearance at end of chemoradiation and at 1 year from end of treatment.

V. To determine the acute and late toxicity rates according to Common Terminology Criteria for Adverse Events (CTCAE) version (v.) 5, including immune-related adverse events (AEs).

VI. To assess patients' quality of life from baseline through 1 year from end of treatment.

EXPLORATORY OBJECTIVES:

I. To determine the overall survival rate at 5-year post-treatment.

II. To determine whether programmed death-ligand 1 (PD-L1) -positive immunohistochemistry and novel quantitative assays correlate to clinical outcome.

III. To determine if the density of infiltrating Cluster of differentiation 3 (CD3)+ T cells/μm2 correlates to clinical outcome.

IV. To monitor immune changes by flow cytometry in the circulating T cell response to EBV antigens.

V. To compare the change in the circulating T-cell repertoire by TCR sequencing and single-cell T-cell profiling.

VI. To quantify treatment-induced changes over time in the circulating T cell immune response to EBV using T-cell receptor (TCR) sequencing and enzyme-linked immunospot (ELISPOT) assays.

OUTLINE:

Patients receive nivolumab intravenously (IV) over 60 minutes on day 1 of courses 1-5 and 7-12. Treatment repeats every 14 days for 11 courses in the absence of disease progression or unacceptable toxicity. Beginning at course 2, patients undergo radiation therapy once daily (QD) 5 days per week and receive cisplatin IV over 30-60 minutes on day 1. Treatment repeats every 7 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 1, 3, 6, 9, and 12 months for up to 1 year and then survival follow-up information may be collected via telephone calls, clinic follow-up visits, or medical records review for up to an additional 4 years. Survival and disease status will be collected until participant death, withdrawal, or if the participant is lost to follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥18 years of age.
2. Histologically or cytologically confirmed nasopharyngeal carcinoma, stage II-IV by American Joint Committee on Cancer (AJCC) 7th edition, endemic-type (defined as World Health Organization (WHO) type 2a and 2b nonkeratinizing or undifferentiated subtypes, excluding WHO type I keratinizing subtype) performed on a biopsy that occurred within 90 days of registration.
3. Positron emission tomography-computed tomography (PET-CT) (preferred) or a CT of chest, abdomen, and pelvis within 60 days of registration showing radiographic stage II to IVB nasopharyngeal cancer.
4. No distant metastasis as verified by one of the study investigators.
5. Documentation that the patient is a candidate for chemoradiation of their nasopharyngeal cancer by one of the study investigators.
6. Ability to tolerate radiation therapy (e.g. lie flat and hold position for treatment).
7. Measurable disease as defined by RECIST v1.1.
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
9. Lack of contraindications to systemic immunotherapy (see list of exclusions below).
10. Resolution of all acute toxic effects of any prior chemotherapy, radiotherapy or surgical procedures to NCI CTCAE Version 5.0 grade 1.
11. Adequate hepatic, hematologic, and renal indices permitting administration of cisplatin and nivolumab (within 14 days of registration):

    Hepatic Function:

    Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 × upper limit of normal (ULN); Total bilirubin ≤ 1.5 × ULN (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL)

    Adequate bone marrow function:

    White blood cells (WBC) ≥ 2000/μL Neutrophils ≥ 1500/μL Platelet ≥ 100 x103/μL Hemoglobin > 9.0 g/dL

    Adequate renal function:

    Serum creatinine ≤ 1.5 × upper limit of normal (ULN) OR

    Creatinine clearance (CrCl) > 40 mL/min (or > 50 mL/min for Singapore sites only) (if using the Cockcroft-Gault formula below):

    Female CrCl = (140 - age in years) x weight in kg x 0.85 72 x serum creatinine in mg/dL Male CrCl = (140 - age in years) x weight in kg x 1.00 72 x serum creatinine in mg/dL
12. Women of childbearing potential must have a negative serum pregnancy test within 24 hours prior to the first dose of study treatment and agree to use appropriate highly effective methods of contraception, during the study and for 5 months following completion of study treatment; A "Woman of childbearing potential" is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal. Menopause is defined clinically as 12 months of amenorrhea in a woman over 45 in the absence of other biological or physiological causes. In addition, women under the age of 62 must have a documented serum follicle stimulating hormone (FSH) level less than 40 milli-international units per milliliter (mIU/mL).

    Female Subjects:

    Women of child bearing potential are expected to use one of the highly effective methods of contraception listed in the protocol.

    Male Subjects:

    Male subjects must inform their female partners who are women of child bearing potential of the contraceptive requirements and are expected to adhere to using contraception with their partner. Female partners of male subjects, who are women of child bearing potential, are expected to use one of the highly effective methods of contraception listed in the protocol. In addition, male subjects are expected to use a condom as noted in the protocol.
13. Men with a female partner of childbearing potential must agree to use highly effective methods of contraception or any contraceptive method with a failure rate of less than 1% per year during the study and for 7 months following completion of study treatment.
14. Ability to sign informed consent.

Exclusion Criteria:

1. Active second malignancy, i.e. patient known to have potentially fatal hematologic malignancy or another solid primary tumor present for which he/she may be (but not necessarily) currently receiving treatment. Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are allowed to enroll in this trial. For example, patients with early-stage skin cancers, prostate cancer under surveillance with non-rising prostate-specific antigen (PSA), or meningioma or thyroid papillary cancers which are under surveillance are eligible. For determinations of a specific clinical condition, please consult with the Principal Investigator.
2. Active, untreated central nervous system (CNS) metastases;
3. Prior treatment with any other anti-programmed cell death protein-1 (anti-PD-1), or PD Ligand-1 (PD-L1) or PD Ligand-2 (PD-L2), anti-cytotoxic T-lymphocyte-associated protein-4 (CTLA-4) antibody, or any other antibody or drug specifically targeting T-cell costimulation or immune checkpoint pathways, or cancer vaccine;
4. Prior systemic cytotoxic therapy, antineoplastic biologic therapy, or major surgery within 28 days of first dose of study medication;
5. Severe hypersensitivity reaction to treatment during prior administration of a monoclonal antibody (mAb) or history of allergy to any study drug component;
6. Has received a live-virus vaccination within 30 days of planned treatment start;
7. Condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration; Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
8. Any evidence of current interstitial lung disease (ILD) or pneumonitis or a prior history of ILD or pneumonitis requiring oral or IV glucocorticoids;
9. Active, known, or suspected autoimmune disease or any autoimmune condition that has required systemic treatment in the past 2 years (replacement therapies for hormone deficiencies are allowed); Subjects are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger.
10. Clinically active diverticulitis, intra-abdominal abscess, gastrointestinal (GI) obstruction, or abdominal carcinomatosis (known risks factors for bowel perforation);
11. Signs or symptoms of infection within 2 weeks prior to first day of study treatment.
12. Patients with active tuberculosis (clinical evaluation in line with local practice), or a known history of active tuberculosis that in the opinion of the treating investigator has a high risk of reactivation.
13. Received therapeutic oral or IV antibiotics within 2 weeks prior to first day of study treatment: Patients receiving prophylactic antibiotics (eg, to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible.
14. Known positive test for human immunodeficiency virus (HIV);
15. Known active hepatitis B or hepatitis C virus (HBV or HCV): Patients with past or resolved HBV infection (defined by a negative hepatitis B surface antigen (HBsAg) test and a positive anti-hepatitis B core antigen (HBc) (anti-HBc)antibody test) are eligible. HBV DNA must be obtained in these patients prior to first day of study treatment. Patients who have been recently discovered to have HBV with positive HBsAg test and positive anti-HBc antibody test but who have been started on antiretroviral treatment with nondetectable HBV DNA are eligible. HBV DNA must be obtained in these patients prior to first day of study treatment
16. Patients with known active hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection: Patients positive for HCV antibody are eligible only if Polymerase chain reaction (PCR) test is negative for HCV RNA.
17. Prior radiation therapy of any type within 7 days of first dose of study medication;
18. Prior radiation therapy to head and neck region that would overlap with intended radiation treatment for nasopharyngeal carcinoma;
19. Medical contraindication to radiation treatment (e.g. active systemic sclerosis, other uncontrolled autoimmune condition)
20. Treatment with prohibited medications (including concurrent anticancer therapy including chemotherapy, radiation, hormonal treatment [except corticosteroids and megestrol acetate] ≤ 14 days prior to treatment.
21. Pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study;
22. Active, uncontrolled psychiatric disorders or substance (drug/alcohol) abuse that interfere with patient's safety, ability to provide informed consent, or ability to comply with the protocol.
23. Persons who are incarcerated or otherwise under compulsory detention by an authority are not eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-02-14 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sue S Yom, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (2):
- University of California, San Francisco, San Francisco, California, United States
- National University Hospital Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Nivolumab + Chemoradiation: Patients receive nivolumab IV over 60 minutes on day 1 of courses 1-5 and 7-12. Treatment repeats every 14 days for 11 courses in the absence of disease progression or unacceptable toxicity. Beginning at course 2, patients undergo radiation therapy once a day (QD) 5 days per week and receive cisplatin IV over 30-60 minutes on day 1. Treatment repeats every 7 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Nivolumab + Chemoradiation
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Nivolumab + Chemoradiation
Number analyzed (Participants) | 40
Age, Customized [Count of Participants; unit: Participants]
  30-39 years old | 3
  40-49 years old | 11
  50-59 years old | 11
  60-69 years old | 13
  70-79 years old | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 38
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 40
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 25
  Singapore | 15

OUTCOME MEASURES:

1. Primary Outcome: Rate of Completion of All Adjuvant Immunotherapy
Description: The rate of completion of all adjuvant therapy by patients treated at the maximum tolerated dose (MTD) schedule will be determined and compared to a historical control rate of 52%, the rate of completion of a standard adjuvant cisplatin-based platform to determine feasibility of study treatment
Time Frame: Up to 1 year
Measure: Number; unit: percentage of participants
Arm/Group | Nivolumab + Chemoradiation
Number analyzed (Participants) | 40
percentage of participants | 100

2. Secondary Outcome: Overall Response Rate (ORR)
Description: The ORR is based on the best overall response (BOR) recorded from the first day of treatment until time of assessment. The percentages of patients with a best overall response rate of complete response (CR), partial response (PR), stable disease (SD), or progressive disease (PD) will be determined as defined by the Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria.
Time Frame: Up to 1 year after completion of treatment
Measure: Number; unit: percentage of participants
Arm/Group | Nivolumab + Chemoradiation
Number analyzed (Participants) | 40
percentage of participants | 100

3. Secondary Outcome: Number of Treatment-related Adverse Events (AEs)
Description: Adverse events will be classified using the National Cancer Institute Common Toxicity Criteria (NCI-CTCAE) version 5.0 by the investigator assessment and reported by frequency of Adverse Events (AEs) attributed as definitely, probably, or possibly related to the study interventions.
Time Frame: Up to 1 year after completion of treatment
Measure: Number; unit: adverse events
Arm/Group | Nivolumab + Chemoradiation
Number analyzed (Participants) | 40
adverse events
  Alanine aminotransferase increased | 1
  Alkaline phosphatase increased | 1
  Allergic rhinitis | 2
  Alopecia | 1
  Anemia | 11
  Anorexia | 18
  Arthralgia | 1
  Bloating | 1
  Blurred vision | 1
  Burn | 1
  Cardiac disorders , Other | 1
  Chills | 4
  Cholesterol high | 1
  Constipation | 14
  Cough | 4
  Dehydration | 7
  Dermatitis radiation | 15
  Diarrhea | 4
  Dizziness | 8
  Dry eye | 1
  Dry mouth | 42
  Dry skin | 3
  Dysgeusia | 42
  Dyspepsia | 1
  Dysphagia | 19
  Dysphasia | 1
  Dyspnea | 1
  Ear and labyrinth disorders, Other | 3
  Ear pain | 2
  Epistaxis | 4
  Eye disorders - Other, specify | 2
  Eye pain | 2
  Fatigue | 30
  Fever | 2
  Gastritis | 1
  Gastroesophageal reflux disease | 1
  Gastrointestinal disorders, Other | 1
  General disorders and administration site conditions - Other, specify | 2
  Gingival pain | 2
  Headache | 5
  Hearing impaired | 10
  Hyperhidrosis | 1
  Hyperkalemia | 2
  Hypermagnesemia | 1
  Hypernatremia | 1
  Hypertension | 1
  Hyperthyroidism | 3
  Hypoalbuminemia | 3
  Hypocalcemia | 4
  Hypokalemia | 8
  Hypomagnesemia | 1
  Hyponatremia | 15
  Hypophosphatemia | 1
  Hypotension | 3
  Hypothyroidism | 7
  Infections and infestations - Other, specify | 2
  Insomnia | 5
  Investigations - Other, specify | 2
  Keratitis | 1
  Lethargy | 1
  Lymph node pain | 1
  Lymphedema | 4
  Lymphocyte count decreased | 38
  Mucositis oral | 43
  Muscle weakness lower limb | 1
  Myalgia | 1
  Nasal congestion | 2
  Nausea | 36
  Neck edema | 2
  Neck pain | 1
  Nervous system disorders, Other | 1
  Neutrophil count decreased | 15
  Non-cardiac chest pain | 1
  Oral pain | 4
  Oropharyngeal pain | 9
  Otitis media | 1
  Pain | 12
  Pain in extremity | 2
  Paresthesia | 3
  Peripheral sensory neuropathy | 5
  Platelet count decreased | 19
  Pruritus | 1
  Psychiatric disorders, Other | 2
  Rash acneiform | 1
  Rash maculo-papular | 1
  Respiratory, thoracic and mediastinal disorders, Other | 2
  Sepsis | 1
  Shingles | 2
  Sinusitis | 4
  Skin and subcutaneous tissue disorders - Other, specify | 25
  Skin hyperpigmentation | 2
  Skin infection | 2
  Skin ulceration | 1
  Sore throat | 10
  Thrush | 10
  Tinnitus | 18
  Tremor | 1
  Urticaria | 2
  Voice alteration | 1
  Vomiting | 7
  Weight loss | 44
  White blood cell decreased | 17

4. Secondary Outcome: Mean Loco-regional Control (LRC) Rate
Description: Duration of LRC will be calculated as 1+ the number of days from the first day of treatment to time of documented locoregional clinical or radiographic relapse, progression or death due to any cause. For patients who continue treatment post-progression, the date of clinical or radiographic relapse or progression will be used for analysis. The Kaplan-Meier analysis will be used to calculate the mean LRC rate with full range.
Time Frame: Up to 1 year after completion of treatment
Measure: Mean (Full Range); unit: days
Arm/Group | Nivolumab + Chemoradiation
Number analyzed (Participants) | 40
days | 96 [89 to 99.6]

5. Secondary Outcome: Mean Distant Metastasis (DM) Rate
Description: Time to DM will be calculated as 1+ the number of days from the first day of treatment to documented clinical or radiographic progression at a distant metastatic site, or death due to any cause. Pathologic confirmation is not required to document the date of distant progression. For patients who continue treatment post-progression, the date of clinical or radiographic progression will be used for analysis. The Kaplan-Meier analysis will be used to calculate the mean DM rate with full range.
Time Frame: Up to 1 year after completion of treatment
Population: As there were no participants with disease progression in a distant metastatic site, no data were collected for this outcome measure.
Measure: Mean (Full Range); unit: days
Arm/Group | Nivolumab + Chemoradiation
Number analyzed (Participants) | 0

6. Secondary Outcome: Mean Change in Scores on the Functional Assessment of Cancer Therapy - Nasopharyngeal Cancer (FACT-NP)
Description: The FACT-NP is a self-report instrument that measures multidimensional quality of life (QOL) in patients with Nasopharyngeal cancer-specific scale. The FACT-NP consists of 43 questions that address physical, social, emotional, and functional well-being, with additional specific questions relevant to persons with nasopharyngeal cancers. Each item has a score range of 0 (Not at all) to 4 (Very much). For the 37 general health and head and neck cancer sections, the raw score range is 0-148, with the higher scores indicating better QOL reported by the participant. The 6 remaining questions for the nasopharyngeal cancers also fall on the same range of 0 to 4, with a raw total score range of 0-24, but on this subscale, lower scores indicate a higher QOL.
Time Frame: Up to 1 year after completion of treatment
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Nivolumab + Chemoradiation
Number analyzed (Participants) | 40
scores on a scale | 3.7 (1.2)

7. Secondary Outcome: Percentage of Participants With Acute Toxicities
Description: Acute toxicity rates will be reported and classified according to CTCAE version 5 and include immune-related AEs
Time Frame: Up to 1 year after completion of treatment
Measure: Number; unit: percentage of participants
Arm/Group | Nivolumab + Chemoradiation
Number analyzed (Participants) | 40
percentage of participants | 100

8. Secondary Outcome: Percentage of Participants With Late Toxicities
Description: Late toxicity rates will be reported and classified according to CTCAE version 5 and include immune-related AEs
Time Frame: Up to 1 year after completion of treatment
Measure: Number; unit: percentage of participants
Arm/Group | Nivolumab + Chemoradiation
Number analyzed (Participants) | 40
percentage of participants | 100

ADVERSE EVENTS:
Time Frame: Up to 1 year after completion of treatment, approximately 18 months
Arm/Group | Nivolumab + Chemoradiation
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 4/40
Other Adverse Events (participants affected / at risk) | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nivolumab + Chemoradiation (N=40)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Hypotension (Vascular disorders) | 2 (2)
Myocardial infarction (Cardiac disorders) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) — Coronavirus disease of 2019 (COVID-19) infection
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nivolumab + Chemoradiation (N=40)
Anemia (Blood and lymphatic system disorders) | 7 (11)
Lymph Node Pain (Blood and lymphatic system disorders) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Cardiac disorders , Other (Cardiac disorders) | 2 (2)
Ear and labyrinth disorders, Other (Ear and labyrinth disorders) | 3 (3)
Ear pain (Ear and labyrinth disorders) | 4 (4)
Hearing impaired (Ear and labyrinth disorders) | 10 (10)
Tinnitus (Ear and labyrinth disorders) | 19 (20)
Hyperthyroidism (Endocrine disorders) | 3 (3)
Hypothyroidism (Endocrine disorders) | 6 (7)
Blurred vision (Eye disorders) | 4 (4)
Dry eye (Eye disorders) | 2 (2)
Eye disorders - Other, specify (Eye disorders) | 4 (5)
Eye pain (Eye disorders) | 2 (2)
Keratitis (Eye disorders) | 1 (1)
Bloating (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 24 (31)
Diarrhea (Gastrointestinal disorders) | 6 (7)
Dry mouth (Gastrointestinal disorders) | 30 (43)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 15 (19)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders, Other (Gastrointestinal disorders) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 28 (45)
Nausea (Gastrointestinal disorders) | 27 (36)
Oral pain (Gastrointestinal disorders) | 3 (4)
Vomiting (Gastrointestinal disorders) | 8 (8)
Chills (General disorders) | 5 (5)
Fatigue (General disorders) | 25 (30)
Fever (General disorders) | 4 (4)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1)
Neck edema (General disorders) | 3 (3)
Non-cardiac chest pain (General disorders) | 2 (2)
Pain (General disorders) | 7 (12)
Allergic Reaction (Immune system disorders) | 1 (1)
Herpes simplex reactivation (Infections and infestations) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 7 (8)
Otitis media (Infections and infestations) | 1 (1)
Papulopustular rash (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Shingles (Infections and infestations) | 3 (3)
Sinusitis (Infections and infestations) | 4 (4)
Skin infection (Infections and infestations) | 1 (2)
Thrush (Infections and infestations) | 11 (12)
Burn (Injury, poisoning and procedural complications) | 1 (1)
Dermatitis radiation (Injury, poisoning and procedural complications) | 16 (16)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (3)
Alkaline phosphatase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 2 (2)
Cholesterol high (Investigations) | 3 (4)
Creatinine increased (Investigations) | 1 (2)
Investigations - Other, specify (Investigations) | 3 (6)
Lymphocyte count decreased (Investigations) | 11 (39)
Neutrophil count decreased (Investigations) | 12 (17)
Platelet count decreased (Investigations) | 11 (21)
Weight loss (Investigations) | 24 (47)
White blood cell decreased (Investigations) | 5 (17)
Anorexia (Metabolism and nutrition disorders) | 15 (18)
Dehydration (Metabolism and nutrition disorders) | 7 (7)
Hyperkalemia (Metabolism and nutrition disorders) | 3 (3)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (5)
Hypokalemia (Metabolism and nutrition disorders) | 3 (9)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 4 (15)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorders, Other (Musculoskeletal and connective tissue disorders) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Anosmia (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 10 (14)
Dysgeusia (Nervous system disorders) | 31 (42)
Dysphasia (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 7 (7)
Lethargy (Nervous system disorders) | 1 (1)
Nervous system disorders, Other (Nervous system disorders) | 2 (2)
Paresthesia (Nervous system disorders) | 3 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 4 (5)
Tremor (Nervous system disorders) | 2 (2)
Depression (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 6 (7)
Psychiatric disorders, Other (Psychiatric disorders) | 2 (2)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 (9)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders, Other (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 9 (10)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (3)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 18 (29)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (2)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (3)
Lymphedema (Vascular disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-12-10): https://cdn.clinicaltrials.gov/large-docs/98/NCT03267498/Prot_SAP_000.pdf